CLINICAL TRIAL: NCT05306574
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, 2-Stage Trial to Evaluate Efficacy and Safety of Telitacicept Compared to Placebo in Patients With Moderately to Severely Active Systemic Lupus Erythematosus (REMESLE-1)
Brief Title: A Study of Telitacicept for the Treatment of Moderately to Severely Active Systemic Lupus Erythematosus (REMESLE-1)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Vor Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC18G001
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telitacicept (Experimental): Telitacicept + Standard of Care (SoC)
  Interventions: Biological: Telitacicept
- Placebo (Placebo Comparator): Placebo + Standard of Care (SoC)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Telitacicept — Subcutaneous injection weekly for 52 weeks
  Other Names: RC18; RC18-L
  Arms: Telitacicept
Biological: Placebo — Subcutaneous injection weekly for 52 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of telitacicept in the treatment of moderately to severely active SLE.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a chronic autoimmune disease with heterogeneous manifestations and disease course. Despite advances in medical care, there are still significant unmet needs in SLE with diminished health-related quality of life (HRQoL), persistent disease activity, disease flares, intolerance to standard of care (SoC) therapies, and development of organ damage and co-morbidities.

Telitacicept is a fully human TACI-Fc fusion protein that targets B lymphocyte stimulator (BLyS) and a proliferating-inducing ligand (APRIL). Blocking the interaction of BLyS and APRIL with their cell membrane receptors (TACI, B-cell maturation antigen (BCMA), and B-cell activating factor receptor (BAFF-R)) would inhibit B cell proliferation and maturation, suppresses immune responses, and may alleviate autoimmune symptoms.

This Phase 3 study is a 2-stage study to evaluate the efficacy and safety of telitacicept compared to placebo in patients with moderately to severely active SLE while receiving SoC treatment in a global patient population with active SLE disease.

* Stage 1: a study to evaluate the efficacy, safety, pharmacokinetics (PK) and PD of two treatment arms of telitacicept compared to placebo in patients with moderately to severely active SLE while receiving SoC treatment.
* Stage 2: a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of telitacicept added to SoC compared to placebo with SoC therapy in patients with moderately to severely active SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-70 years at screening.
2. Has a diagnosis of SLE for at least 6 months prior to the screening visit.
3. Meets the 2019 EULAR/ACR Classification criteria for SLE.
4. Moderately to severely active SLE defined by the following:

   1. SELENA SLEDAI total score ≥6 points with clinical SLEDAI score ≥4 points at screening;
   2. BILAG organ system scores of at least 1A or 2B at screening.
5. Clinical SLEDAI score of ≥4 at Day 0 prior to randomization.
6. At least one positive serologic parameter within the screening period.
7. Currently receiving at least one of the SOC SLE medications: oral corticosteroid, antimalarial and/or immunosuppressive agent.

Exclusion Criteria:

1. Active lupus nephritis undergoing induction therapy or unstable renal diseases within 12 weeks prior to screening.
2. Active or unstable neuropsychiatric SLE.
3. Autoimmune or rheumatic disease other than SLE

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
SLE Responder Index (SRI-4) | Week 52
  Proportion of subjects achieving an SLE Responder Index (SRI-4) response at Week 52

SECONDARY OUTCOMES:
SLE Responder Index (SRI-4) | Week 24
  Proportion of subjects achieving an SLE Responder Index (SRI-4) response at Week 24
Achieve and sustain a low dose of corticosteriods | Weeks 52
  Proportion of subjects achieving the target of corticosteroids reduction through Week 52.
SLE Responder Index (SRI-4) and sustaining a low dose of corticosteriods | Week 52
  Proportion of patients achieving an SRI-4 response at Week 52, while achieving and maintaining corticosteroids reduction.
BILAG-based Combined Lupus Assessment (BICLA) Response | Week 52
  Proportion of patients achieving a BILAG-based Combined Lupus Assessment (BICLA) response at Week 52
Time to Flare | Week 52
  Time to flare assessed by SELENA-SLEDAI Flare Index (SFI) from baseline through Week 52
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Week 52
  Proportion of patients achieving clinically meaningful improvement in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) at Week 52

CONTACTS AND LOCATIONS:
Locations (77):
- United States (12):
  - Anniston, Alabama Site, Anniston, Alabama
  - Mission Hills Site, Mission Hills, California
  - Orange Site, Orange, California
  - Thousands Oaks Site, Thousand Oaks, California
  - Miami, FL Site, Miami, Florida
  - Tampa, Florida Site, Tampa, Florida
  - Wheaton, Maryland Site, Wheaton, Maryland
  - Grand Blanc Site, Grand Blanc, Michigan
  - Baytown Site, Baytown, Texas
  - Colleyville, Texas Site, Colleyville, Texas
  - Houston Site, Houston, Texas
  - Waco Site, Waco, Texas
- Argentina (7):
  - Quilmes Site, Quilmes, Buenos Aires
  - Rosario Site, Rosario, Santa Fe Province
  - San Miguel de Tucuman Site 1, San Miguel de Tucumán, Tucumán Province
  - San Miguel de Tucuman Site 2, San Miguel de Tucumán, Tucumán Province
  - Ciudad Autonoma Buenos Aires Site 2, Ciudad Autonoma Buenos Aires
  - Cordoba Site, Córdoba
  - San Juan Site, San Juan
- Australia (2):
  - Garran Site, Garran, Austl. Cap. Terr.
  - Murdoch Site, Murdoch, Western Australia
- Bulgaria (9):
  - Pleven Site, Pleven
  - Plovdiv Site, Plovdiv
  - Ruse Site, Rousse
  - Sevlievo Site, Sevlievo
  - Sofia Site 1, Sofia
  - Sofia Site 4, Sofia
  - Sofia Site 5, Sofia
  - Sofia Site 3, Sofia
  - Stara Zagora Site, Stara Zagora
- Chile (4):
  - Santiago Site 4, Santiago
  - Santiago Site 1, Santiago
  - Santiago Site 3, Santiago
  - Santiago Site 2, Santiago
- Colombia (5):
  - Barranquilla site, Barranquilla
  - Bucaramanga site, Bucaramanga
  - Medellin Site 1, Medellín
  - Medellin site 2, Medellín
  - Monteria site, Montería
- Germany (2):
  - Koeln Site, Cologne, North Rhine-Westphalia
  - Muenster Site, Münster, North Rhine-Westphalia
- Guatemala site, Guatemala City, Guatemala
- Hungary (3):
  - Budapest Site, Budapest
  - Debrecen Site, Debrecen
  - Gyula Site, Gyula
- Quatre Bornes Site, Quatre Bornes, Mauritius
- Mexico (5):
  - Cuernavaca Site, Cuernavaca
  - Guadalajara Site, Guadalajara
  - Ciudad de Mexico Site, Mexico City
  - Mexico site 1, México
  - Mexico Site 2, México
- Philippines (5):
  - Batangas Site, Batangas
  - Cagayan de Oro City Site, Cagayan de Oro
  - Los Baños Site, Los Baños
  - Makati City Site, Makati City
  - Manila Site, Manila
- Poland (16):
  - Bydgoszcz Site, Bydgoszcz
  - Bydgoszcz Site 2, Bydgoszcz
  - Bydgoszcz Site 3, Bydgoszcz
  - Bytom Site, Bytom
  - Katowice Site, Katowice
  - Krakow Site 1, Krakow
  - Lodz Site, Lodz
  - Malbork Site, Malbork
  - Poznan Site 2, Poznan
  - Poznan SIte, Poznan
  - Poznań Site, Poznan
  - Szczecin Site, Szczecin
  - Warszawa Site 2, Warsaw
  - Warszawa Site 3, Warsaw
  - Warszawa Site, Warsaw
  - Wroclaw Site 2, Wroclaw
- Puerto Rico (2):
  - Caguas Site, Caguas
  - San Juan Site, San Juan
- Spain (3):
  - Sevilla Site 1, Seville
  - Sevilla Site 2, Seville
  - Valencia Site, Valencia

IPD SHARING:
Plan to Share IPD: No